CLINICAL TRIAL: NCT02186041
Title: Sacral Neuromodulation With InterStim® Therapy for Intractable Urinary Voiding Dysfunctions (SOUNDS):an Observational Study
Brief Title: Sacral Neuromodulation With InterStim® Therapy for Intractable Urinary Voiding Dysfunctions (SOUNDS): an Observational Study
Acronym: SOUNDS
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Collaborators: Medtronic France SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: 1.05.7008
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Urinary Incontinence; Over Active Bladder; Urinary Retention
MeSH Terms: conditions — Urinary Incontinence; Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- De-Novo patients: Patients tested and de novo implanted with Interstim®. These patients will be followed-up for 5 years after the implant visit.
  Interventions: Device: Sacral Nerve Modulation
- Device replacement: Patients implanted with Interstim® for a device replacement. These patients will be followed-up for 5 years after the implant visit.
  Interventions: Device: Sacral Nerve Modulation
- Not-implanted patients: Patients who are tested and are not implanted with the Interstim® system. The data of the follow up of the test will be captured up to one year after the end-test visit
  Interventions: Device: Sacral Nerve Modulation

INTERVENTIONS:
Device: Sacral Nerve Modulation
  Other Names: Interstim

SUMMARY:
The purpose of this study is to document the safety, the effectiveness, the continued performance at mid and long term, the morbidity and the percent of surgical revisions of the Interstim® therapy for up to 5 years in a representative sample of French centers under real-life conditions of use.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old;
* Patient signed the Patient Data Release Form;
* Patient suffering from retention or Over Active Bladder;
* Patient is eligible for Interstim® system therapy.

Exclusion Criteria:

* Difficulty of collecting follow up patient data;
* Patient not affiliated to social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are eligible for Interstim® therapy for the treatment of intractable urinary voiding dysfunctions will be proposed to participate to the registry in a representative selection of French centers.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Safety and Performance (2 years) - Objective #1 | 24 months
  To evaluate the safety of Interstim® therapy and the performance of the Interstim® system in the 2 years following the enrollment.
  The rate of surgical revisions/explantations of the Interstim® system or any of its parts will be measured.

SECONDARY OUTCOMES:
Safety and Performance (5 years) - Objective #2 | 5 years
  To evaluate the safety of Interstim® therapy and the performance of the Interstim® system in the 5 years following the enrollment.
  The rate of adverse device events and device deficiencies will be measured.
Concomitant treatment - Objective #3 | Up to 5 years
  To evaluate the use of concomitant treatments or interventions dedicated to intractable urinary voiding dysfunctions.
NRS evaluation - Objective#4 | Up to 5 years
  To evaluate the effect of InterStim® therapy on the perceived bother resulting from conditions as measured on Numeric Rating Scale (NRS) up to 5 years follow up.
Effect of Therapy in UR patients - Objective #5 | Up to 5 years
  To assess the effect of Interstim® therapy on the subset of patients with urinary retention as measured by the number of self-catheterizations per day.
Effect of therapy on OAB patients - Objective#6 | Up to 5 years
  To assess the effect of Interstim® therapy on the subset of patients with Over Active Bladder (OAB wet and OAB dry) symptom as measured by the number of voids and leaks per day.
Quality of Life (DITROVIE) - Objective#7 | Up to 5 years
  To assess the therapy effect on Quality of Life using the DITROVIE questionnaire.
Quality of Life (EQ-5D-5L) - Objective#8 | Up to 5 years
  To assess the therapy effect on Quality of Life using the EQ-5D-5L questionnaire.
Urinary symptoms (USP) - Objective#9 | Up to 5 years
  To evaluate the change of urinary symptoms of all patients implanted with Interstim® using the Urinary Symptom Profile (USP) questionnaire.
Goal attainment assessment - Objective#10 | Up to 5 years
  To evaluate the long term goal attainment assessed by the GAS.
Assessment of Fecal Incontinence - Objective#11 | Up to 5 years
  To assess the therapy effect on fecal incontinence for subset of patients with double incontinence using the WEXNER fecal incontinence score.

CONTACTS AND LOCATIONS:
Locations (24):
- France (24):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - CHIC Alencon Mamers, Alençon
  - CHU Angers, Angers
  - Hopital Prive Sevigné, Cesson Sevigné
  - Clinique Chirurgicale du Pre, Le Mans
  - CHRU Lille, Lille
  - Clinique Mutualiste de la porte de l'Orient, Lorient
  - Clinique Mutualiste de la Porte de lOrient, Lorient
  - APM Hopital de La Conception, Marseille
  - APHM Hôpital Nord, Marseille
  - Hopital Robert Schuman, Metz
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - CHU Bordeaux - Centre Universitaire Pellegrin, Pessac
  - Maison des consultations - Centre Briochin d'Urologie, Plérin
  - Groupe Courlancy, Reims
  - CH Roubaix, Roubaix
  - CHU Rouen - Hopital Charles Nicolle, Rouen
  - Clinique Urologique Nantes Atlantis, Saint-Herblain
  - CH Sarreguemines, Sarreguemines
  - Hopital Civil Strasbourg, Strasbourg
  - Polyclinique Ormeau, Tarbes
  - CHU Toulouse - Hopital Rangueil, Toulouse
  - Clinique Ambroise Pare, Toulouse

REFERENCES:
- [Derived] Chartier-Kastler E, Normand LL, Ruffion A, Saussine C, Braguet R, Rabut B, Ragni E, Perrouin-Verbe MA, Pierrevelcin J, Rousseau T, Game X, Tanneau Y, Dargent F, Biardeau X, Graziana JP, Stoica G, Brassart E, Fourmarier M, Yaghi N, Capon G, Ferchaud J, Berrogain N, Peyrat L, Pecoux F, Bryckaert PE, Melotti A, Abouihia A, Keller DUJ, Cornu JN. Sacral Neuromodulation with the InterStim System for Overactive Bladder: 3-Year Results from the French Prospective, Multicenter, Observational SOUNDS Study. Eur Urol Focus. 2022 Sep;8(5):1399-1407. doi: 10.1016/j.euf.2021.06.013. Epub 2021 Jul 30. PMID 34334342
- [Derived] Chartier-Kastler E, Le Normand L, Ruffion A, Dargent F, Braguet R, Saussine C, Tanneau Y, Graziana JP, Ragni E, Rabut B, Rousseau T, Biardeau X, Game X, Pierrevelcin J, Brassart E, Fourmarier M, Stoica G, Berrogain N, Yaghi N, Pecoux F, Capon G, Ferchaud J, Peyrat L, Bryckaert PE, Karsenty G, Melotti A, Abouihia A, Keller DUJ, Cornu JN. Sacral Neuromodulation with the InterStim System for Intractable Lower Urinary Tract Dysfunctions (SOUNDS): Results of Clinical Effectiveness, Quality of Life, Patient-Reported Outcomes and Safety in a French Multicenter Observational Study. Eur Urol Focus. 2021 Nov;7(6):1430-1437. doi: 10.1016/j.euf.2020.06.026. Epub 2020 Sep 7. PMID 32907782